CLINICAL TRIAL: NCT00046475
Title: A Multi-Center, Double-Blind, Randomized, Placebo-Controlled, Crossover Study to Assess the Clinical Benefit of Midodrine Hydrochloride in Patients With Neurogenic Orthostatic Hypotension
Brief Title: A Study for Patients With Neurogenic Orthostatic Hypotension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 20,762-401
Record Dates: First submitted 2002-09-30; First posted 2002-10-02 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Hypotension, Orthostatic
MeSH Terms: conditions — Hypotension, Orthostatic | interventions — Midodrine

INTERVENTIONS:
Drug: Midodrine Hydrochloride

SUMMARY:
We are seeking male and female patients to voluntarily take part in a clinical research study. Patients must be aged 18 or older and diagnosed with symptomatic orthostatic hypotension (low blood pressure while in the upright position) due to Parkinson's disease, multiple system atrophy, pure autonomic failure or autonomic neuropathies (i.e. neurogenic orthostatic hypotension). Symptoms of low blood pressure include dizziness, lightheadedness, changes in vision and generalized weakness upon standing. The main effect of the drug being studied is to increase blood pressure in the upright position so symptoms will decrease.

The purpose of this clinical study is to further assess the clinical benefit of midodrine hydrochloride (ProAmatine®), an approved treatment for orthostatic hypotension. During the course of the study, participants will receive either ProAmatine® or a placebo. Assessments will be made using questionnaires that measure symptom and activity levels. Blood pressure in the lying down and standing positions will be measured at each visit.

ELIGIBILITY:
Inclusion Criteria:

* The male or female patient must be 18 years of age or older and ambulatory.
* Female patients must be: without menses for at least 12 months prior to screening; surgically sterilized (bilateral tubal ligation or hysterectomy); or practicing adequate means of birth control. Adequate means of birth control is defined as the use of prescribed birth control pills, IUD, or hormonal injections from at least one month prior to screening. Double-barrier methods and abstinence are also acceptable forms of birth control.
* The patient has been diagnosed with symptomatic orthostatic hypotension due to Parkinson's disease, multiple system atrophy, pure autonomic failure or autonomic neuropathies (i.e. neurogenic orthostatic hypotension).
* The patient manifests at least one of the following symptoms while standing or has a history of one of the following when not treated for orthostatic hypotension: dizziness, lightheadedness, feeling faint or feeling like they may black out.
* The patient is willing and able to undergo the procedures required by this protocol including morning office visits, assessment completion, protocol compliance and participation in the wash-out period.
* The patient signs an Institutional-Review-Board approved written Informed Consent form prior to any study procedures taking place.

Exclusion Criteria:

* The patient is pregnant or lactating female.
* The patient has pre-existing sustained supine hypertension greater than 180 systolic and 110 diastolic mmHg.
* The patient is taking medications such as vasodilators, pressors, diuretics, ACE inhibitors, angiotensin receptor blockers, beta-blockers, combined alpha and beta-blockers, MAOI's, herbals, or specific mixed effect medications.
* The Principal Investigator deems any laboratory test abnormality clinically significant.
* The patient has a diagnosis of any of the following disorders at the time of screening: pheochromocytoma; cardiac conditions including: congestive heart failure within the previous 6 months, myocardial infarction within the previous 6 months, symptomatic coronary artery disease, history of ventricular tachycardia, or uncontrolled cardiac arrhythmias; thyrotoxicosis; uncontrolled diabetes mellitus (uncontrolled defined as HgbA1c greater than or equal to 10%); history of cerebrovascular accident, transient ischemic attack (TIA) or symptomatic carotid artery stenosis within the previous 6 months; history of coagulopathies; pulmonary hypertension; severe psychiatric disorders; renal failure (creatinine equal to or greater than 2 times the upper limit of normal).
* The patient has a concurrent chronic or acute illness, disability, or other condition that might confound the results of the tests and/or measurements administered in this trial, or that might increase the risk to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 1997-12-01 (Actual); Primary Completion 1999-11-24 (Actual); Study Completion 1999-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (15):
- United States (15):
  - North Alabama Neuroscience Research, Huntsville, Alabama
  - Dr. Harry Pepe & Associates, Inc., Miramar, Florida
  - Suncoast Neuroscience Associates, Inc., St. Petersburg, Florida
  - Economou & Associates, LTD, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Michigan Pain and Neurological Institute, Ann Arbor, Michigan
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - NY Presbyterian Hospital, New York, New York
  - Medical College of Ohio, Toledo, Ohio
  - COR Clinical Research, LLC, Oklahoma City, Oklahoma
  - Westmoreland Neurology Associates Inc., Greensburg, Pennsylvania
  - Neurological Associates of Delaware Valley, Upland, Pennsylvania
  - Diabetes & Glandular Disease Research Associates, PA, San Antonio, Texas
  - Monarch Medical Research, Norfolk, Virginia
  - West Virginia University, Morgantown, West Virginia

REFERENCES:
- See also: The National Dysautonomia Research Foundation — http://www.ndrf.org
- See also: Clinical Trials Resource Site — http://www.centerwatch.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients who completed the Titration Period were then randomized to receive either Midodrine/Placebo or Placebo/Midodrine during Treatment Periods 1 and 2. Some patients did not meet the criteria for randomization, had an AE, or withdrew from the study after completing the Titration Period prior to entering Treatment Period 1.
Groups:
- All Enrolled Participants: All patients who were enrolled in this study are included in this population.
- Midodrine/Placebo: Participants received their optimum dose of Midodrine HCl for 2 weeks, followed by 2 weeks of treatment with Placebo
- Placebo/Midodrine: Participants received Placebo for 2 weeks, followed by 2 weeks of treatment with their optimum dose of Midodrine HCl
Period: Screening/Washout Period (Up to 2 Weeks)
Arm/Group | All Enrolled Participants | Midodrine/Placebo | Placebo/Midodrine
Started | 140 | 0 | 0
Completed | 136 | 0 | 0
Not Completed | 4 | 0 | 0
Period: Titration (1 Week)
Arm/Group | All Enrolled Participants | Midodrine/Placebo | Placebo/Midodrine
Started | 136 | 0 | 0
Completed | 136 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Treatment Period 1 (Up to 2 Weeks)
Arm/Group | All Enrolled Participants | Midodrine/Placebo | Placebo/Midodrine
Started | 0 | 45 (Patients did not meet the criteria for randomization, had an AE, or withdrew from the study.) | 60 (Patients did not meet the criteria for randomization, had an AE, or withdrew from the study.)
Completed | 0 | 45 | 59
Not Completed | 0 | 0 | 1
Period: Treatment Period 2 (Up to 2 Weeks)
Arm/Group | All Enrolled Participants | Midodrine/Placebo | Placebo/Midodrine
Started | 0 | 45 | 59
Completed | 0 | 44 | 59
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population, defined as all patients who were randomly assigned to treatment in the study and have at least one post-randomization Orthostatic Hypotension Questionnaire (OHQ) measurement.
Groups:
- Total: Total of all reporting groups
Arm/Group | Midodrine/Placebo | Placebo/Midodrine | Total
Number analyzed (Participants) | 45 | 59 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (14.22) | 62.2 (14.43) | 62.2 (14.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 22 | 35 | 57

OUTCOME MEASURES:

1. Primary Outcome: Post-treatment Score For Item 1 of The Orthostatic Hypotension Symptom Assessment (OHSA) Scale
Description: Item 1 of the OHSA asked the patient to rate, using a 0-10 scale (0 meaning not bothered and 10 meaning the worst), his or her impression of the severity of dizziness, lightheadedness, feeling faint, or feeling like you might black out whenever he or she was standing and that improved when he or she sat or laid down. Higher scores indicate more severe disease.
Time Frame: End of 2-week treatment period
Population: Intent-to-Treat, defined as all patients who were randomly assigned to treatment in the study and have at least one post-randomization OHQ measurement.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Midodrine HCl: Participants received their optimum dose (5-50mg) of Midodrine HCl for 2 weeks
- Placebo: Participants received Placebo daily for 2 weeks
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 103 | 103
scores on a scale | 4.1 (2.9) | 5.2 (2.7)
Statistical Analysis 1: Comparison: Midodrine HCl vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA — The P-value is based on an ANOVA model with post-treatment responses for OHSA Item 1 as dependent variable, treatment, sequence, period (Visit 5 or 6), as fixed effects, and patient within sequence as random effect

2. Primary Outcome: Re-analysis of The Post-treatment Score For Item 1 of The OHSA Scale, Excluding Two Sites
Description: as for outcome 1
Time Frame: End of 2-week treatment period
Population: Intent-to-Treat, defined as all patients who were randomly assigned to treatment in the study and have at least one post-randomization OHQ measurement. Data for 2 sites were excluded from this re-analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 94 | 94
scores on a scale | 4.3 (2.93) | 5.1 (2.76)
Statistical Analysis 1: Comparison: Midodrine HCl vs Placebo; Test type: Superiority or Other; p = 0.011, ANOVA — The P-value is based on an ANOVA model with post-treatment responses for OHSA Item as dependent variable, treatment, sequence, period (Visit 5 or 6), as fixed effects, and patient within sequence as random effect

3. Secondary Outcome: Change From Baseline in The OHSA Items 2 Through 6 Scores
Description: Items 2 through 6 of the OHSA asked the patient to rate, using a 0-10 scale (0 meaning not bothered and 10 meaning the worst), his or her impression of the severity of the following symptoms whenever he or she was standing and that improved when he or she sat down or laid down: Item 2 addresses problems with vision (blurring, seeing spots, tunnel vision, etc); Item 3, weakness; Item 4, fatigue; Item 5, trouble concentrating; and Item 6, head or neck discomfort. Symptomatology was assessed at Visit 3A (titration), Visit 5 (Period 2), and Visit 6 (study completion). A negative change from baseline indicates that symptoms have improved.
Time Frame: From the time of titration until the end of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 103 | 103
scores on a scale
  Item 2, n= 103, 103 | -1.2 (2.5) | -0.2 (2.3)
  Item 3, n=103, 103 | -1.3 (3.2) | -0.4 (2.5)
  Item 4, n=103, 103 | -1.2 (3.2) | -0.4 (2.6)
  Item 5, n=102, 102 | -0.4 (2.7) | 0.0 (2.2)
  Item 6, n=102, 102 | -0.8 (2.6) | -0.5 (2.1)
Statistical Analysis 1: Comparison: Midodrine HCl vs Placebo; Analysis of Item 2; Test type: Superiority or Other; p < 0.001, ANOVA — The P-value is based on an ANOVA model with post-treatment responses for OHSA Item 2 as dependent variable, treatment, sequence, period (Visit 5 or 6), as fixed effects, and patient within sequence as random effect
Statistical Analysis 2: Comparison: Midodrine HCl vs Placebo; Analysis of Item 3; Test type: Superiority or Other; p = 0.002, ANOVA — The P-value is based on an ANOVA model with post-treatment responses for OHSA Item 3 as dependent variable, treatment, sequence, period (Visit 5 or 6), as fixed effects, and patient within sequence as random effect
Statistical Analysis 3: Comparison: Midodrine HCl vs Placebo; Analysis of Item 4; Test type: Superiority or Other; p = 0.004, ANOVA — The P-value is based on an ANOVA model with post-treatment responses for OHSA Item 4 as dependent variable, treatment, sequence, period (Visit 5 or 6), as fixed effects, and patient within sequence as random effect
Statistical Analysis 4: Comparison: Midodrine HCl vs Placebo; Analysis of Item 5; Test type: Superiority or Other; p = 0.026, ANOVA — The P-value is based on an ANOVA model with post-treatment responses for OHSA Item 5 as dependent variable, treatment, sequence, period (Visit 5 or 6), as fixed effects, and patient within sequence as random effect
Statistical Analysis 5: Comparison: Midodrine HCl vs Placebo; Analysis of Item 6; Test type: Superiority or Other; p = 0.226, ANOVA — The P-value is based on an ANOVA model with post-treatment responses for OHSA Item 6 as dependent variable, treatment, sequence, period (Visit 5 or 6), as fixed effects, and patient within sequence as random effect

4. Secondary Outcome: Change From Baseline in The OHSA Composite Symptom Score
Description: The OHSA composite symptom score was calculated by taking the average of the ratings for the symptoms present at Baseline. Participants were asked to rate symptoms by using a 0-10 scale (0 meaning not bothered and 10 meaning the worst). For subsequent visits, only those symptoms present at Baseline were scored. In this manner, a score was produced that represents the severity (and subsequent change in severity) of the patient's neurogenic OH symptoms, regardless of how many symptoms are presented at Baseline. Symptomatology was assessed at Visit 3A (titration), Visit 5 (Period 2), and Visit 6 (study completion). A negative change from baseline indicates that symptoms have improved.
Time Frame: From the time of titration until the end of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 102 | 102
scores on a scale | -1.3 (2.5) | -0.54 (1.952)
Statistical Analysis 1: Comparison: Midodrine HCl vs Placebo; Test type: Superiority or Other; p = 0.002, ANOVA — The P-value is based on an ANOVA model with post-treatment composite symptom score as dependent variable, treatment, sequence, period (Visit 5 or 6), as fixed effects, and patient within sequence as random effect

5. Secondary Outcome: Change From Baseline in The Orthostatic Hypotension Daily Activity Scale (OHDAS) Items 1 Through 4 Scores
Description: The OHDAS had 4 items that asked the patient to give a graduated score from 0 (no limitation due to OH) to 10 (complete limitation due to OH). Item 1 addressed activities that required standing for a short time; Item 2, activities that required standing for a long time; Item 3, activities that required walking for a short time; and Item 4, activities that required walking for a long time. Symptomatology was assessed at Visit 3A (titration), Visit 5 (Period 2), and Visit 6 (study completion). A negative change from baseline indicates that symptoms have improved.
Time Frame: From the time of titration until the end of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 104 | 104
scores on a scale
  Item 1, n=102, 101 | -1.1 (2.90) | -0.4 (1.95)
  Item 2, n=98, 99 | -1.8 (3.14) | -0.6 (2.41)
  Item 3, n=100, 101 | -1.1 (2.71) | -0.2 (2.16)
  Item 4, n=89, 90 | -1.3 (3.31) | -0.5 (2.57)
Statistical Analysis 1: Comparison: Midodrine HCl vs Placebo; Analysis of Item 1; Test type: Superiority or Other; p < 0.001, ANOVA — The P-value is based on an ANOVA model with post-treatment responses for OHDAS Item 1 as dependent variable, treatment, sequence, period (Visit 5 or 6), as fixed effects, and patient within sequence as random effect
Statistical Analysis 2: Comparison: Midodrine HCl vs Placebo; Analysis of Item 2; Test type: Superiority or Other; p < 0.001, ANOVA — The P-value is based on an ANOVA model with post-treatment responses for OHDAS Item 2 as dependent variable, treatment, sequence, period (Visit 5 or 6), as fixed effects, and patient within sequence as random effect
Statistical Analysis 3: Comparison: Midodrine HCl vs Placebo; Analysis of Item 3; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is based on an ANOVA model with post-treatment responses for OHDAS Item 3 as dependent variable, treatment, sequence, period (Visit 5 or 6), as fixed effects, and patient within sequence as random effect
Statistical Analysis 4: Comparison: Midodrine HCl vs Placebo; Analysis of Item 4; Test type: Superiority or Other; p = 0.001, ANOVA — The P-value is based on an ANOVA model with post-treatment responses for OHDAS Item 4 as dependent variable, treatment, sequence, period (Visit 5 or 6), as fixed effects, and patient within sequence as random effect

6. Secondary Outcome: Change From Baseline in The Orthostatic Hypotension Global Daily Activity Score
Description: The OHDAS global daily activity score was calculated as the average of all daily activity item scores. The OHDAS had 4 items that asked the patient to give a graduated score from 0 (no limitation due to OH) to 10 (complete limitation due to OH) to activities that required standing for a short time, standing for a long time, walking for a short time, walking for a long time. Symptomatology was assessed at Visit 3A (titration), Visit 5 (Period 2), and Visit 6 (study completion). A negative change from baseline indicates that symptoms have improved.
Time Frame: From the time of titration until the end of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 103 | 103
scores on a scale | -1.4 (2.6) | -0.4 (1.9)
Statistical Analysis 1: Comparison: Midodrine HCl vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA — The P-value is based on an ANOVA model with post-treatment global daily activity score as dependent variable, treatment, sequence, period (Visit 5 or 6), as fixed effects, and patient within sequence as random effect

7. Secondary Outcome: Percent of Participants Scored as Improved on The Clinician Version of The Clinical Global Impressions Improvement (CGI-I) Scale
Description: The CGI-I is a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Clinical Global Impressions ratings are completed with respect to neurogenic OH symptoms. A value of 0 was used if the investigator or patient assessment was not performed. The improved category is made up of patients who were evaluated as very much improved, much improved, or slightly improved for the classification of "Overall Improvement." The CGI-I was completed at Visit 5 (Period 2) and Visit 6 (study completion).
Time Frame: From the time of titration until the end of treatment
Population: as for outcome 1
Measure: Number; unit: percent of participants
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 104 | 104
percent of participants | 73.1 | 45.2

8. Secondary Outcome: Percent of Participants Scored as Improved on The Patient Version of The CGI-I Scale
Description: as for outcome 7
Time Frame: From the time of titration until the end of treatment
Population: as for outcome 1
Measure: Number; unit: percent of participants
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 104 | 104
percent of participants | 62.5 | 50.0

9. Secondary Outcome: Change From Baseline in Standing Blood Pressure (BP)
Description: Standing BP was measured at Visit 5 (Period 2) and Visit 6 (study completion) and compared to measurements taken at Visit 3A (titration). Standing BP was measured 3 minutes after the patient rose from the supine position or as soon as the patient indicated they needed to sit down. If the patient indicated he or she needed to sit down, the BP measurement was taken while in the standing position, before the patient sat down.
Time Frame: From the time of titration until the end of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 104 | 104
mmHg
  Systolic Pressure | 10.7 (21.68) | 2.8 (19.55)
  Diastolic Pressure | 5.9 (14.46) | 1.5 (13.03)
Statistical Analysis 1: Comparison: Midodrine HCl vs Placebo; Analysis of standing systolic blood pressure; Test type: Superiority or Other; p = 0.002, ANOVA — The P-value is based on an ANOVA model with change from baseline standing systolic blood pressure as dependent variable, treatment, sequence, period (Visit 5 or 6), as fixed effects, and patient within sequence as random effect
Statistical Analysis 2: Comparison: Midodrine HCl vs Placebo; Analysis of standing diastolic blood pressure; Test type: Superiority or Other; p = 0.010, ANOVA — The P-value is based on an ANOVA model with change from baseline standing diastolic blood pressure as dependent variable, treatment, sequence, period (Visit 5 or 6), as fixed effects, and patient within sequence as random effect

10. Secondary Outcome: Change From Baseline in Supine BP
Description: Supine BP was measured at Visit 5 (Period 2) and Visit 6 (study completion) and compared to measurements taken at Visit 3A (titration). Supine BP was measured after the patient had been in the supine position for 5 minutes.
Time Frame: From the time of titration until the end of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 104 | 104
mmHg
  Systolic Pressure | 7.6 (22.76) | -0.9 (15.74)
  Diastolic Pressure | 3.4 (11.89) | 0.3 (10.35)
Statistical Analysis 1: Comparison: Midodrine HCl vs Placebo; Analysis of supine systolic blood pressure; Test type: Superiority or Other; p < 0.001, ANOVA — The P-value is based on an ANOVA model with change from baseline supine systolic blood pressure as dependent variable, treatment, sequence, period (Visit 5 or 6), as fixed effects, and patient within sequence as random effect
Statistical Analysis 2: Comparison: Midodrine HCl vs Placebo; Analysis of supine diastolic blood pressure; Test type: Superiority or Other; p = 0.002, ANOVA — The P-value is based on an ANOVA model with change from baseline supine diastolic blood pressure as dependent variable, treatment, sequence, period (Visit 5 or 6), as fixed effects, and patient within sequence as random effect

11. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Version 2 Health Survey Questionnaire Scores
Description: The SF-36 consists of 36 items in eight domains: physical functioning, general health, role-physical, bodily pain, vitality, social functioning, role-emotional, and mental health. Version 2 references "one week ago" for some questions. Raw scale scores for the SF-36 were transformed to a 0-100 scale with a higher score indicating a better quality of life. A positive change from baseline indicates that symptoms have improved. The SF-36 was completed at Visit 5 (Period 2) and Visit 6 (study completion) and compared to the score from Visit 3A (titration).
Time Frame: From the time of titration until the end of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 70 | 69
scores on a scale
  General Health | 1.97 (7.801) | 1.59 (6.027)
  Physical Functioning | 1.99 (8.255) | 1.71 (8.034)
Statistical Analysis 1: Comparison: Midodrine HCl vs Placebo; Analysis of general health; Test type: Superiority or Other; p = 0.569, ANOVA — The P-value is based on an ANOVA model with SF-36 general health score as dependent variable, treatment, sequence, period (Visit 5 or 6), as fixed effects, and patient within sequence as random effect
Statistical Analysis 2: Comparison: Midodrine HCl vs Placebo; Analysis of physical functioning; Test type: Superiority or Other; p = 0.578, ANOVA — The P-value is based on an ANOVA model with SF-36 physical functioning score as dependent variable, treatment, sequence, period (Visit 5 or 6), as fixed effects, and patient within sequence as random effect

12. Secondary Outcome: Test Reliability of the Intent-to-Treat (ITT) Population
Description: Item 1 of the OHSA, the OHSA composite score, and the OHDAS global daily activity score were analyzed for test-retest reliability as a measure of validity. Test-retest reliability is the Pearson product-moment correlation coefficient calculated between OHQ scores at Visit 3A (baseline measure) and OHQ scores at Visit 5 for the subjects who received Placebo during Randomization Period 1.
Time Frame: From the time of titration until the end of treatment
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Groups:
- ITT Population: All patients who were randomly assigned to treatment in the study and have at least one post-randomization OHQ measurement.
Arm/Group | ITT Population
Number analyzed (Participants) | 59
correlation coefficient
  OHSA Item 1 | 0.53
  OHSA Composite Score | 0.61
  OHDAS Global Daily Activity Score | 0.66

13. Secondary Outcome: Responsiveness of the Intent-to-Treat (ITT) Population
Description: Item 1 of the OHSA, the OHSA composite score, and the OHDAS global daily activity score were analyzed for responsiveness as a measure of validity. Assuming that subjects who received Placebo during Randomization Period 1 are stable between Visit 3A and Visit 5, and using them as the stable subjects, responsiveness was calculated as [(OH CFB in Midodrine group)-(OH CFB in Placebo group)]/(SD of OH CFB in Placebo group), where CFB is change from baseline, SD is the standard deviation of OH CFB of the stable subjects; the value reported is the quotient of this equation.
Time Frame: From the time of titration until the end of treatment
Population: as for outcome 1
Measure: Number; unit: quotient
Arm/Group | ITT Population
Number analyzed (Participants) | 59
quotient
  OHSA Item 1 | -0.4099
  OHSA Composite Score | -0.4014
  OHDAS Global Daily Activity Score | -0.4903

14. Secondary Outcome: Convergent Validity of the Intent-to-Treat (ITT) Population
Description: Item 1 of the OHSA and the OHSA composite score were analyzed for convergent validity with the CGI-I-Clinician scores. The change from baseline in the CGI-I scores are correlated with the OHSA Item 1 score change from baseline and the OHSA composite score change from baseline for the subjects in the ITT population. Values shown are Spearman correlation coefficients.
Time Frame: From the time of titration until the end of treatment
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Arm/Group | ITT Population
Number analyzed (Participants) | 104
correlation coefficient
  OHSA Item 1, n=103 | 0.36
  OHSA Composite Score, n=102 | 0.38

15. Primary Outcome: Post-treatment OHSA Item 1 Score of United States (US) Participants With Mild/Moderate Disease According to The Clinical Global Impressions-Severity (CGI-S) Scale
Description: Item 1 of the OHSA asked the patient to rate, using a 0-10 scale (0 meaning not bothered and 10 meaning the worst), his or her impression of the severity of dizziness, lightheadedness, feeling faint, or feeling like you might black out whenever he or she was standing and that improved when he or she sat or laid down. The results are reported by degree of severity according to the CGI-S scale, which uses 4 categories to describe disease severity: Mild, Moderate, Marked, and Severe. The Item 1 scores reported are grouped for participants with Mild or Moderate disease severity. Higher scores indicate more severe disease.
Time Frame: End of 2-week treatment period
Population: Randomized participants enrolled at any of the 28 US sites
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 39 | 39
scores on a scale | 4.4 (2.97) | 3.8 (2.63)
Statistical Analysis 1: Comparison: Midodrine HCl vs Placebo; Analysis of US participants with mild or moderate disease severity; Test type: Superiority or Other; p = 0.370, ANOVA — The p-value is based on an ANOVA model with post-treatment responses for OHSA Item 1 as dependent variable, treatment, sequence, period (Visit 5 or 6), as fixed effects, and subject-within sequence as random effect

16. Primary Outcome: Post-treatment OHSA Item 1 Score of US Participants With Marked/Severe Disease According to The CGI-S Scale
Description: Item 1 of the OHSA asked the patient to rate, using a 0-10 scale (0 meaning not bothered and 10 meaning the worst), his or her impression of the severity of dizziness, lightheadedness, feeling faint, or feeling like you might black out whenever he or she was standing and that improved when he or she sat or laid down. The results are reported by degree of severity according to the CGI-S scale, which uses 4 categories to describe disease severity: Mild, Moderate, Marked, and Severe. The Item 1 scores reported are grouped for participants with Marked or Severe disease severity. Higher scores indicate more severe disease.
Time Frame: End of 2-week treatment period
Population: Randomized participants enrolled at any of the 28 US sites
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 30 | 30
scores on a scale | 4.7 (2.90) | 6.1 (2.60)
Statistical Analysis 1: Comparison: Midodrine HCl vs Placebo; Analysis of US participants with marked or severe disease severity; Test type: Superiority or Other; p = 0.007, ANOVA — [p-value comment as in outcome 15, analysis 1]

ADVERSE EVENTS:
Groups:
- Screening/Washout: Patients signed the informed consent form and were screened for eligibility. Eligible patients were off drug for 1 week.
- Titration: Patients received different doses of drug for at least 2 weeks to determine the maximum tolerated dose.
- Midodrine HCl: Patients received their optimum dose of Midodrine HCl for 2 weeks.
- Placebo: Patients received Placebo for 2 weeks.
- Follow-up: Patients were contacted 30 days after last study drug dose to follow up on any ongoing AEs and inquire if there were any new AEs.
Arm/Group | Screening/Washout | Titration | Midodrine HCl | Placebo | Follow-up
Serious Adverse Events (participants affected / at risk) | 1/140 | 4/136 | 0/104 | 1/105 | 5/140
Other Adverse Events (participants affected / at risk) | 12/140 | 42/136 | 22/104 | 23/105 | 23/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Screening/Washout (N=140) | Titration (N=136) | Midodrine HCl (N=104) | Placebo (N=105) | Follow-up (N=140)
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Blindness cortical (Eye disorders) | 0 | 1 | 0 | 0 | 0
Colitis NOS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage NOS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Injury NOS (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Therapeutic agent poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Convulsions NOS (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Parkinson's disease NOS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Screening/Washout (N=140) | Titration (N=136) | Midodrine HCl (N=104) | Placebo (N=105) | Follow-up (N=140)
Urinary tract infection NOS (Infections and infestations) | 5 | 6 | 1 | 1 | 7
Dizziness (Nervous system disorders) | 3 | 7 | 3 | 5 | 5
Headache NOS (Nervous system disorders) | 1 | 13 | 6 | 7 | 5
Paraesthesia (Nervous system disorders) | 0 | 10 | 5 | 5 | 3
Pruritus NOS (Skin and subcutaneous tissue disorders) | 0 | 11 | 8 | 8 | 9
Hypertension NOS (Vascular disorders) | 4 | 9 | 3 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.